CLINICAL TRIAL: NCT01085513
Title: Intestinal Motility Evaluation by Endoluminal Image Analysis Using Capsule Endoscopy (CE-EIA): a Multi-center Clinical Trial
Brief Title: Diagnosis of Intestinal Motility by Image Analysis Using Capsule Endoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MA-68
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-01

CONDITIONS: Intestinal Abnormalities
Keywords: intestinal abnormalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Active Comparator): Patients previously indicated for manometry
  Interventions: Device: PillCam SB2
- Healthy volunteers (Active Comparator): Healthy volunteers
  Interventions: Device: PillCam SB2

INTERVENTIONS:
Device: PillCam SB2 — The disposable, ingestible PillCam SB 2 Capsule, part no. FGS-0180, is designed to acquire video images during natural propulsion through the small bowel. The capsule transmits acquired images via RF communication channel to the DataRecorder located outside the body.

SUMMARY:
Conventional intestinal manometry is the current gold standard for the evaluation of intestinal motility, and identifies patterns of intestinal dysmotility. However intestinal manometry involves intestinal intubation with consequent discomfort for the patients, and requires considerable technical expertise and knowledge for interpretation of the data. Hence, to date this method has limited indications and is restricted to very few referral centers around the world.

A novel method for evaluation of intestinal motility has been developed based on endoluminal image analysis using the endoscopic PillCam capsule, In contrast to manometry, this technique is minimally invasive, the technical aspects are simple, and the analysis is fully automated by a computer program.

The technique has been validated in a group of patients with intestinal dysmotility and healthy subjects, and has demonstrated over 90% sensitivity and specificity.

This technique needs now to be validated in a large multinational population, to further develop a robust discrimination algorithm for widespread diagnostic application. Furthermore, whereas manometry only recognizes neuropathic, myopathic and obstructive motor patterns, endoluminal image analysis may identify different categories of patients depending on the clinical presentation and the etiologic factors involved.

This study is designed to provide evidence that the algorithm, using images created by PillCam SB2 capsules, is at least as good as small bowel manometry in diagnosing severe dysmotility.

DETAILED DESCRIPTION:
Conventional intestinal manometry is the current gold standard for the evaluation of intestinal motility1,2,3,11, and identifies patterns of intestinal dysmotility4,8,9. However intestinal manometry involves intestinal intubation with consequent discomfort for the patients. Furthermore, it requires considerable technical expertise and knowledge for interpretation of the data. Hence, to date this method has limited indications and is restricted to very few referral centers around the world6,7,10,13.

Vall d'Hebron Hospital, in collaboration with CVC (Barcelona, Spain) have recently developed a minimally invasive method for evaluation of intestinal motility based on endoluminal image analysis using the endoscopic PillCam capsule. In contrast to manometry, this technique is minimally invasive, the technical aspects are simple, and the analysis is performed fully automated by a computer program. Both the technical procedure of the test and the endoluminal image analysis program has been developed by a multidisciplinary medical-engineering team in the Autonomous University of Barcelona over the past 5 years. The technique has been validated in a group of patients with intestinal dysmotility and healthy subjects, and has demonstrated over 90% sensitivity and specificity.

In brief, the technique works as follows. In each study a series of features are analyzed: contractile patterns (contractions evaluated as a diaphragmatic occlusion of the lumen and by the presence of a radial wrinkle pattern), non contractile patterns (wall and tunnel patterns), luminal content (turbid pattern), endoluminal motion, and capsule displacement.

The program is based on an automated learning method (machine learning technique). Data from patients and healthy subjects are used as a training set. Based on these data, the program develops the function that best discriminates both groups. The performance of the system has been validated using the leave-one-out method that uses all but one as training set and evaluates the left-out example.

This technique needs now to be validated in a large multinational population. Using this expanded pool of studies as a learning set, a robust discrimination algorithm will be developed, that can be made available for widespread diagnostic application. Furthermore, whereas manometry only recognizes neuropathic, myopathic5,12 and obstructive motor patterns, endoluminal image analysis may identify different categories of patients depending on the clinical presentation and the etiologic factors involved.

This study is designed to provide evidence that the algorithm, using images created by PillCam SB2 capsules, is at least as good as small bowel manometry in diagnosing severe dysmotility.

ELIGIBILITY:
Inclusion criteria - Patients

* Patient's age is 16-80 years, inclusive.
* One of the following SB manometry procedures:

  * Underwent SB manometry within five years if results were abnormal
  * Underwent SB manometry within 1 year if results were normal
  * Scheduled for SB manometry within six months of enrollment date
* Patient was indicated for small bowel manometry based on one or both of the following symptoms:

  * Pseudo obstruction of the small bowel: symptoms resembling mechanical small bowel obstruction without evidence of luminal compromise of the gut. Mechanical occlusion is ruled-out by endoscopic and / or radiological studies following the criteria of the attending physician.

Patients may have any of the following:

* recurrent acute episodes (at least two) with air fluid levels (as evidenced at least once by abdominal X-ray), or
* chronic symptoms with small bowel dilation resembling a partial mechanical obstruction.

Patients will be tested during period of (non-acute) remission. - Chronic severe GI symptoms with inability to maintain normal body weight: abdominal symptoms (such as nausea, abdominal distension, discomfort or pain) produce inability to maintain a normal body weight as defined by unintentional weight loss of at least 10% of original body weight before onset of symptoms or a BMI < 18.5, while on a normal diet (without oral dietary supplements, enteral or parenteral feeding).

These should be chronic symptoms lasting at least 6 months.

- Patient or legal guardian agrees to sign consent form

Exclusion criteria - Patients

* Acute exacerbation of chronic obstructive symptoms.
* Mechanical obstruction of any kind such as definite long stricture seen on radiological exam.
* Suspected GI stricture, followed by Agile® study that could not prove patency of the GI tract.
* Known history of small bowel organic disease such as Crohn's Disease or Celiac.
* Patient suffers from any condition, such as swallowing problems or having an implanted cardiac pacemaker or defibrillator which precludes compliance with study and/or device instructions.
* Non-steroidal anti-inflammatory drugs including aspirin, (twice weekly or more) during the 4 weeks preceding the CE exam.
* Patient has undergone gastrectomy (segmental small bowel resection over 30%).
* During the period between small bowel manometry and Capsule endoscopy, the patient has undergone any abdominal surgical procedures other than appendectomy, cholecystectomy, abdominal wall hernia repair or catheter placing for enteral feeding.
* Manometry was performed before any other allowed GI procedure.
* Patient is pregnant.
* Known abuse of alcohol or illicit substances.
* Patient presently presenting with an acute life threatening condition.
* Participating in another clinical study within 30 days.

Inclusion criteria - Healthy Volunteers

* Volunteer's age is 16-80 years, inclusive.
* Volunteer or legal guardian agrees to sign consent form. 6.5.2 Exclusion criteria - Healthy Volunteers
* Known diabetes mellitus
* Recurrent Gastrointestinal symptoms
* Volunteer suffers from any condition, such as swallowing problems, which precludes compliance with study and/or device instructions
* Non-steroidal anti-inflammatory drugs including aspirin, (twice weekly or more) during the 4 weeks preceding enrollment
* More than one answer above 'mild' on the healthy volunteer symptoms questionnaire (Appendix C).
* Female volunteer is pregnant
* Known abuse of alcohol or illicit substances.
* Participating in another clinical study within 30 days

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Azpiroz, Prof., Principal Investigator — Universitat Autonoma de Barcelona
Locations (6):
- United States (2):
  - Division of Gastroenterology and Hepatology Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic,, Rochester, Minnesota
- Center for GI Research, KU Leuven,, Leuven, Belgium
- Internal Medicine & Gastroenterology, University of Bologna,, Bologna, Italy
- Autonomous University of Barcelona, Barcelona, Spain
- Departement of Internal Medicine, Sahlgrenska Universitetss, Gothenburg, Sweden

RESULTS

PARTICIPANT FLOW:
Period: Phase I - Development Phase
Arm/Group | Patients | Healthy Volunteers
Started | 54 | 52
Completed | 54 (recruitment was premature terminated) | 52
Not Completed | 0 | 0
Period: Phase II - Validation Phase
Arm/Group | Patients | Healthy Volunteers
Started | 21 | 16
Completed | 21 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: no analysis has been performd since study was premature terminated
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients | Healthy Volunteers | Total
Number analyzed (Participants) | 75 | 68 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (15.34) | 40.5 (13.6) | 40.34 (14.49)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 68 | 64 | 132
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 43 | 96
  Male | 22 | 25 | 47
Region of Enrollment [Number; unit: participants]
  United States | 7 | 0 | 7
  Belgium | 14 | 16 | 30
  Spain | 37 | 47 | 84
  Italy | 16 | 3 | 19
  Sweden | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Accuracy of Endoluminal Image Analysis by Capsule Endoscopy in Detecting Severe Dysmotility
Description: Patients were indicated for small bowel manometry based on one or both of the following symptoms:
  * Pseudo obstruction
  * Unintentional body weight loss
Time Frame: Up to 7 months
Population: Total of 143 cases were enrolled. Phase 1- total of 106 cases (52 healthy volunteers, 54 patients) provided sensitivity and specificity results to train an algorithm.
  Phase 2- total of 37 cases (16 healthy volunteers, 21 patients) was intended to validate the sensitivity/specificity but study was terminated and the 37 cases were not analyzed.
Measure: Number; unit: percentage
Arm/Group | Healthy Volunteers | Patients
Number analyzed (Participants) | 52 | 54
percentage
  Sensitivity | 90 | 90
  Specificity | 100 | 100

2. Secondary Outcome: To Assess Correlation Between Patient Clinical Symptoms and CE-EIA
Description: The study was terminated without achieving the needed sample size due to very low recruitment rate. Therefore, no statistical analysis has been performed to achieve the secondary outcome.
Time Frame: Up to 7 months
Population: The 2ndary outcome was to be calculated from subjects in Phase 2 (i.e. the validation phase) of the study but the study was terminated and the 37 participants in phase 2 were not analyzed
Arm/Group | Healthy Volunteers | Patients
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AE information was collected as occurs from screening visit through follow up phone call which could occur over up to 7 months
Groups:
- Patients: Patients previously indicated for manometry
  Two Moderate adverse events not related to studies procedure were reported within this study: abdominal pain and nausea.
  In one case (i.e., abdominal pain) emergency visit occurred and the adverse events was resolved within four days.
Arm/Group | Patients | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/68
Other Adverse Events (participants affected / at risk) | 2/75 | 0/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients (N=75) | Healthy Volunteers (N=68)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study terminated early due to slow recruitment. Phase 1 of the study enrolled but was intended to train an algorithm only.The validation phase 2 which supported objectives was not completed and the study objectives could not be evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No